CLINICAL TRIAL: NCT05342714
Title: Safety and Efficacy of Remote Ischemic Conditioning in Patients With Chronic Cerebral Artery Occlusion: A Prospective, Randomized, Controlled Study
Brief Title: Remote Ischemic Conditioning for Chronic Cerebral Artery Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIC-CCAO
Record Dates: First submitted 2022-03-30; First posted 2022-04-25 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Artery Occlusion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): Participants in the experimental group receive both RIC and standard clinical therapy. The RIC treatment is composed of 5 cycles of bilateral upper limb ischemia for 5 minutes followed by reperfusion for another 5 minutes performed twice a day for a total of 180 consecutive days.The procedure was performed by using an electric autocontrol device with cuffs that inflated to a pressure of 200 mmHg during the ischemic period and deflated during the reperfusion (Patent No.CN200820123637.X, China).
  Interventions: Device: Remote ischemic conditioning
- Control group (No Intervention): Participants in the control group receive standard clinical therapy.

INTERVENTIONS:
Device: Remote ischemic conditioning — The LRIC treatment consisted of 5 cycles of bilateral upper limb ischemia for 5 minutes followed by reperfusion for another 5 minutes performed twice a day for a total of 180 consecutive days.The procedure was performed by using an electric autocontrol device with cuffs that inflated to a pressure of 200 mmHg during the ischemic period and deflated during the reperfusion.(Patent No.CN200820123637.X, China).
  Arms: RIC group

SUMMARY:
Chronic cerebral artery occlusion (CCAO), which is characterized by the pathophysiological change of long-term cerebral hemodynamic disorder, is one of the major risk factors affect the occurrence and recurrence of ischemic stroke. However, the mechanism of CCAO injury is not clear and effective treatment is warranted. The purpose of this study is to investigate the protective effect and underlying mechanism of remote ischemic conditioning (RIC) on CCAO.

DETAILED DESCRIPTION:
CCAO is a cerebrovascular disease due to cerebral hypo-perfusion. It is often associated with repeated ischemic stroke or transient neurological symptoms, progressive cognitive decline and reduction of daily ability. Specific and effective treatment is warranted for symptomatic management of CCAO. RIC is a non-invasive strategy to protect the brain. The clinical trials have demonstrated that daily limb RIC seems to be potentially effective in patients with symptomatic intracranial arterial stenosis in cerebral blood flow and metabolism. RIC can also ameliorate cerebral small vessel disease in slowing cognition decline and reducing white matter. Therefore, it is worth to investigate the neuroprotective mechanism of RIC for CCAO.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age range 40-80 years, regardless of gender;
* (2) Digital angiography (DSA) / ultrasound / CT angiography (CTA) / magnetic resonance angiography (MRA) showed unilateral internal carotid artery (ICA) or middle cerebral artery (MCA) occlusion and stenosis of any other cerebral arteries (e.g. the other side of ICA or MCA, basilar artery) < 50%;
* (3) Modified Rankin Scale (mRS) score 0-2;
* (4) Symptoms of ischemic cerebrovascular disease (ischemic stroke or TIA) due to ICA or MCA occlusions within 12 months prior to enrollment;
* (5) neurological deficits were stable ≥ 30 days after occlusion;
* (6) Magnetic resonance perfusion weighted imaging (PWI) showed mean transit time (MTT) ≥ 4s and related cerebral blood flow (rCBF) (symptomatic side/asymptomatic side) < 0.95;
* (7) The subject or its legally authorized representative is able to provide informed reports.

Exclusion Criteria:

* (1) Uncontrolled hypertension despite the use of antihypertensive drugs before enrollment (defined as systolic blood pressure ≥200mmHg);
* (2) Stenosis or occlusion of subclavian artery and upper limb artery;
* (3) Previous history of cerebral hemorrhage, including intracranial hemorrhage, ischemic stroke hemorrhage transformation, vascular malformation or intracranial tumor or other parts of the active bleeding disease;
* (4) History of brain tumor or mental illness or acute stroke ≤6 months;
* (5) Suffering from cardiogenic thrombosis diseases, such as mitral stenosis and atrial fibrillation, myocardial infarction, mural thrombosis or valvular vegetations, congestive heart failure or endocarditis within six months;
* (6) Obvious disorder of coagulation mechanism;
* (7) Severe liver or kidney insufficiency, malignant tumor, or serious diseases requiring medical intervention or surgery;
* (8) There is soft tissue or blood vessel injury at the cuff compression site of RIC treatment, or other conditions that cannot tolerate RIC;
* (9) Pregnant or lactating women;
* (10) Life expectancy <6 months;
* (11) Refusal to sign informed consent, poor compliance, or inability to complete complete treatment, etc.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of cerebral blood flow perfusion | 180 days
  The investigators evaluate the change of perfusion capacity of cerebral blood vessels on PWI-MRI.

SECONDARY OUTCOMES:
Recurrence times of stroke or transient ischemic attack (TIA) | 180 days
  The investigators evaluate the times of stroke or transient ischemic attack (TIA) recurrence.
Changes of volume of WMHs | 180 days
  The investigators evaluate the the change of volume of WMHs on Flairs-MRI.
Change of the direction of white matter cellulose | 180 days
  The investigators evaluate the change of direction of white matter cellulose on DTI-MRI.
Change of cerebral hemoglobin oxygenation status | 180 days
  The investigators evaluate the change of cerebral hemoglobin oxygenation status on BOLD-rsfMRI.
Change of collateral circulation | 180 days
  The investigators evaluate the change of collateral circulation on ASL-MRI.
Change of the Montreal Cognitive Assessment (MoCA) score | 180 days
  The investigators evaluate the change of neurobehavioral function by the Montreal Cognitive Assessment (MoCA) score. The minimum value is 0 and maximum value is 30. The higher scores represent the better outcome.
Change of the Verbal Fluency Test (VFT) score | 180 days
  The investigators evaluate the change of neurobehavioral function by the Verbal Fluency Test (VFT) score. The minimum value is 0 and without the maximum value. The higher scores represent the better outcome.
Change of the Digit Span Forward and Backward score | 180 days
  The investigators evaluate the change of neurobehavioral function by the Digit Span Forward and Backward score. The minimum value is 3 and maximum value is 12. The higher scores represent the better outcome.
Change of the Hamilton Depression-17 (HAMD-17) scale | 180 days
  The investigators evaluate the change of neuropsychological function by the Hamilton Depression-17 (HAMD-17) scale. The minimum value is 0 and maximum value is 54. The higher scores represent the worse outcome.
Change of the Hamilton Anxiety (HAMA) scale | 180 days
  The investigators evaluate the change of neuropsychological function by the Hamilton Anxiety (HAMA) scale. The minimum value is 0 and maximum value is 56. The higher scores represent the worse outcome.
Adverse events related to RIC treatment | From baseline to 180-day treatment
  Adverse events related to RIC treatment, such as mucocutaneous hemorrhage, changes in coagulation function and so on.

OTHER OUTCOMES:
Safety of RIC [Number of patients not tolerating RIC procedure and patients with erythema or skin lesions related to RIC] | 180 days
  The safety of RIC by the number of patients not tolerating RIC procedure and patients with erythema or skin lesions related to RIC.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD.PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meng R, Asmaro K, Meng L, Liu Y, Ma C, Xi C, Li G, Ren C, Luo Y, Ling F, Jia J, Hua Y, Wang X, Ding Y, Lo EH, Ji X. Upper limb ischemic preconditioning prevents recurrent stroke in intracranial arterial stenosis. Neurology. 2012 Oct 30;79(18):1853-61. doi: 10.1212/WNL.0b013e318271f76a. Epub 2012 Oct 3. PMID 23035060
- [Result] Wang Y, Meng R, Song H, Liu G, Hua Y, Cui D, Zheng L, Feng W, Liebeskind DS, Fisher M, Ji X. Remote Ischemic Conditioning May Improve Outcomes of Patients With Cerebral Small-Vessel Disease. Stroke. 2017 Nov;48(11):3064-3072. doi: 10.1161/STROKEAHA.117.017691. Epub 2017 Oct 17. PMID 29042490